CLINICAL TRIAL: NCT03226964
Title: Assessment of High Flow Nasal Cannula Oxygenation in EBUS Bronchoscopy
Acronym: AHOE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Hospital Galway (Other)
Responsible Party: Principal Investigator, Mohammed Ahmed, Specialist Registrar in Respiratory Medicine, University College Hospital Galway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.0
Record Dates: First submitted 2017-03-14; First posted 2017-07-24 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Lung Cancer; Lymphadenopathy
Keywords: endobronchial ultrasound; high flow nasal oxygen
MeSH Terms: conditions — Lung Neoplasms; Lymphadenopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High flow nasal oxygen (Experimental): (Optiflow; Fisher & Paykel, Auckland, New Zealand)
  Interventions: Device: high flow nasal oxygen
- Nasal prongs (Active Comparator)
  Interventions: Device: high flow nasal oxygen

INTERVENTIONS:
Device: high flow nasal oxygen — humidified high flow nasal oxygen

SUMMARY:
This study is a prospective randomised trial where a computer will randomly allocate

patients to one of two possible methods of delivering oxygen during the procedure of

bronchoscopy. This trial compares high flow nasal cannula (HFNC) with nasal prongs in

delivering oxygen to patients undergoing endo-bronchial ultrasound guided trans-

bronchial nodal aspiration (EBUS-TBNA) a specialised form of bronchoscopy procedure.

HFNC uses humidified higher gas flow rates than conventional low flow systems such as

nasal prongs which are limited by the respiratory rate and effort.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a peripheral arterial pulse oximetry ≥ 90% breathing room air
* Age ≥ 18 years
* Able to breathe spontaneously throughout the procedure

Exclusion Criteria:

* Respiratory or cardiac failure
* Recent myocardial infarction < 6 weeks ago
* On long term oxygen therapy, those with tracheostomy and/ or non-invasive or invasive mechanical ventilation
* Nasal and/ or nasopharyngeal disease
* Inability to give informed consent
* Dementia
* Hepatic or end stage renal disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
drop in oxygen saturation during procedure | through procedure completion defined as withdrawing scope from patient's mouth, an average of 30 minutes
  the difference in oxygen saturation levels between pre-treatment assessments and the lowest saturation level achieved during treatment

SECONDARY OUTCOMES:
change in venous CO2 | 1 hour after procedure
  Change in venous CO2 1 hour after procedure compared to pre-procedure level
end tidal CO2 during procedure | through procedure completion defined as withdrawing scope from patient's mouth an average of 30 minutes
  Measured with tip of scope at lower trachea
Patient experience measure on a visual analogue scale | up to 3 hours after procedure
endotracheal intubation during or post procedure | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: David Breen, Study Chair — University Hospital Galway
Locations (1):
- University Hospital Galway, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No